CLINICAL TRIAL: NCT02941224
Title: SELUTION™ Sirolimus Coated PTA Balloon Catheter Prospective, Controlled, Multi-Center, Open, Single-Arm Clinical Investigation for the Treatment of Patients With Femoropopliteal Artery Lesions With a Novel Drug Coated Balloon
Brief Title: First-in-human Evaluation of the SELUTION DCB, a Novel Sirolimus Coated Balloon in Peripheral Arteries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-1001
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Patients With Peripheral Artery Disease in the SFA or PA

ARMS (1):
- SELUTION DCB (Experimental): The SELUTION™ DCB (coated with sirolimus) is intended for use as a Percutaneous Transluminal Angioplasty (PTA) balloon catheter to dilate de-novo or restenotic vascular lesions, for the purpose of improving limb perfusion and decreasing the incidence of restenosis.
  Interventions: Device: SELUTION DCB (sirolimus coated balloon)

INTERVENTIONS:
Device: SELUTION DCB (sirolimus coated balloon)

SUMMARY:
The primary objective of the Clinical Investigation is to assess the clinical safety and the inhibition of restenosis of the Investigational Device in the treatment of de-novo occluded/stenotic or re-occluded/restenotic lesions of the superficial femoral and/or popliteal arteries.

The primary endpoint of the Clinical Investigation is Late Lumen Loss (LLL) of the target lesion, as measured by Quantitative Vascular Angiography (QVA) at 6 months post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are mentally and linguistically able to understand the aim of the Clinical Investigation and to show sufficient compliance in following the Clinical Investigation Plan.
2. Patients must agree to return for all required post-index procedure follow-up visits.
3. Patients are able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of the Clinical Investigation. Patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.
4. Patients have a documented diagnosis of Peripheral Arterial Disease (PAD) classified as Rutherford class 2-3-4 in the Superficial Femoral Artery (SFA) and/or Popliteal Artery (PA). Patients with a documented diagnosis of PAD classified as Rutherford class 2, may only be included in case conservative and medicinal treatment have proved ineffective in these patients.
5. Patients are able to walk without assistive devices such as walker or cane.
6. Patients are eligible for peripheral revascularization by means of PTA.
7. The target vessel reference diameter must be ≥ 3.0 and ≤ 7.0 mm.
8. The target lesion length must be ≤ 15 cm and stenosed or occluded.
9. The target lesion must be in a native, non-stented SFA and/or PA target vessel and located ≥ 1 cm below the Common Femoral Artery (CFA) bifurcation and terminate distally ≥ 1 cm above the origin of the Tibial-Peroneal (TP) trunk.
10. Treatment of multiple target lesions is allowed, as long as the composite target lesion length is ≤ 15 cm and the target lesions can be treated with a maximum of 2 overlapping Investigational Devices.
11. The target lesion must either be de-novo or restenotic (stenosis ≥ 70% diameter reduction or occlusion by visual estimate). If the target lesion is restenotic, the prior PTA must have been done > 30 days prior-index procedure.
12. The target lesion must have been successfully crossed with a guide wire and there must be successful pre-dilatation of the target lesion, in the absence of early recoil, significant remaining stenosis or flow-limiting dissection.
13. There must be a patent (< 50% stenosis) inflow artery, as confirmed by angiography. Treatment of inflow disease during the index procedure is allowed. Patients with flow-limiting inflow lesions can be included, if inflow lesions have been treated (use of DES or DCB not allowed) successfully (attainment of residual diameter stenosis ≤ 30% without major vascular complications).

There must be at least 1 patent (< 50% stenosis) native outflow artery to the ankle, as confirmed by angiography. Treatment of outflow disease during the index procedure is NOT permitted.

Exclusion Criteria:

1. Patients with a known hypersensitivity or contraindication to aspirin, heparin, other anticoagulant/anti-platelet therapies, Sirolimus (or analogs) or sensitivity to contrast media that cannot be adequately pre-medicated.
2. Patients with an obligatory need of cumarine or other anticoagulants (e.g. Novel Oral Anticoagulant (NOAC) drugs).
3. Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the Investigational Device.
4. Patients with a life expectancy, from the Investigator's opinion, of less than 3 years.
5. Patients that are currently participating in other clinical investigations involving any investigational drug or device that may potentially confound the results of the Clinical Investigation, or that would limit the patient's compliance with the follow-up requirements of the Clinical Investigation.
6. Patients with a history of Myocardial Infarction (MI), thrombolysis or angina within 30 days prior-index procedure.
7. Patients with a history of major disabling stroke within 3 months prior-index procedure.
8. Patients with any type of previous or planned surgical or interventional procedure within 15 days prior- and/or within 30 days post-index procedure.
9. Patients with a presence or history of severe renal failure (Glomerular Filtration Rate (GFR) ≤ 30 ml/min).
10. Patients who have undergone prior vascular surgery of the SFA and/or PA in the index limb to treat atherosclerotic disease.
11. Patients with clinically significant aneurysmal disease of the iliac, femoral or popliteal artery and patients with a history of clinically significant abdominal aortic aneurysm.
12. Treatment of the contralateral limb during the same index procedure or within 30 days post-index procedure in order to avoid confounding complications.
13. Patients under administrative or judicial custody (§20 Act on Medical Devices, Germany).
14. Composite target lesion length is > 15 cm.
15. Treatment of target lesion(s) that requires more than 2 overlapping Investigational Devices.
16. A COMPLIANCE360-Score of 3 or higher, showing a (moderately) severe circumferentially calcified target lesion as displayed on plain x-ray prior to the index procedure expected for early recoil and imperative need of plaque modulation or stenting as judged by the investigator prior to pre-dilatation.
17. Significant inflow disease or treatment of inflow disease during index procedure not successful.
18. Known inadequate distal outflow (> 50 % stenosis of distal popliteal and/or all three tibial vessels), or planned treatment of vascular disease distal to the target lesion post-index procedure.
19. Known required use of adjunctive treatment modalities (laser, atherectomy, cryoplasty, scoring/cutting balloon, etc.).

Remaining acute or sub-acute thrombus in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) of the target lesion, as measured by Quantitative Vascular Angiography (QVA) | 6 Months (plus or minus 30 days)

SECONDARY OUTCOMES:
Device success | index procedure
  defined as successful delivery, inflation, deflation and retrieval of the Investigational Device
Procedural success | index procedure
  defined as final residual stenosis of ≤ 30% of the target lesion, as measured by QVA
Clinical success | within 24 hours post-index procedure
  defined as procedural success with no MAE noted
Freedom from device- and procedure- related death | 30 days
Freedom from Major Adverse Event (MAE) | 6 Months (plus or minus 30 days)
  defined as composite rate of Cardio-Vascular (CV) mortality, index limb amputation, target lesion thrombosis and clinically driven Target Lesion Revascularization (TLR)
Primary Patency (PP) | discharge, 6, 12 and 24 Months (plus or minus 30 days)
  defined as freedom from clinically driven Target Lesion Revascularization (TLR) and freedom from restenosis as determined by Duplex Ultrasound (DUS) with a Peak Systolic Velocity Ratio (PSVR) < 2.5 of the target lesion
Composite of freedom from index limb amputation and clinically driven Target Vessel Revascularization (TVR) | 12 and 24 Months (plus or minus 30 days)
Angiographic Binary Restenosis (ABR) | 6 Month (plus or minus 30 days)
  defined as > 50% diameter stenosis of the target lesion, as measured by QVA
Change of Rutherford Classification as compared to baseline | at 6, 12 and 24 months (plus or minus 30 days)
Change of Ankle Brachial Index (ABI) as compared to baseline | at 6, 12 and 24 months (plus or minus 30 days)
Change in functional status measured by changes in the Walking Impairment compared to baseline | at 6, 12 and 24 months (plus or minus 30 days)
Change in functional status measured by changes in the general health-related Quality of Life measured by changes in EQ-5D-5L questionnaire compared to baseline | at 6, 12 and 24 months (plus or minus 30 days)
User Acceptance Testing (UAT) questionnaire | index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof Dr Med, Principal Investigator — Universitäts-Herzzentrum Freiburg-Bad Krozingen
Locations (4):
- Germany (4):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Radiologische Gemeinschaftspraxis Ihre-Radiologen Franziskus - Krankenhaus Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Evangelisches Krankenhaus Hubertus, Berlin

REFERENCES:
- [Derived] Zeller T, Brechtel K, Meyer DR, Noory E, Beschorner U, Albrecht T. Six-Month Outcomes From the First-in-Human, Single-Arm SELUTION Sustained-Limus-Release Drug-Eluting Balloon Trial in Femoropopliteal Lesions. J Endovasc Ther. 2020 Oct;27(5):683-690. doi: 10.1177/1526602820941811. Epub 2020 Jul 15. PMID 32666871